CLINICAL TRIAL: NCT06312891
Title: Value of Heart Rate Lowering Therapy in Acute Myocarditis
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mahmoud Moustafa, Resident at student hospital , assiut university, Assiut University
Other Study IDs: VOHRLTIAM
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis | interventions — Ivabradine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional anti-inflammatory treatment (control group).
- Conventional ttt PLUS Carvedilol.
- Conventional ttt PLUS Ivabradine.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — heart rate lowering therapy
  Groups: Conventional ttt PLUS Ivabradine.

SUMMARY:
To study the value of heart rate lowering therapy "pharmacological rest" on the short term in cases of myocarditis without LV dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adults: ≥18 years of age.
* Presentation: at least one of the following:

  * Myopericarditis/ACS-like
  * MINOCA
  * Arrhythmias: brady or tachyarrhythmias.
  * Unexplained compensated acute cardiomyopathy (excluded ischemic, valvular, hypertensive, metabolic, and toxic causes of cardiomyopathy as indicated clinically).
* TTE: LVEF>40%
* CMR-confirmed myo(peri)carditis (Lake Louise criteria)

Exclusion Criteria:

* • Rheumatic carditis.

  * Connective tissue diseases (-ve ANA).
  * Cancer chemotherapy.
  * Toxicity from immunotherapy.
  * Vaccine-related myocarditis.
  * Presence of coronary artery disease.
  * Peripartum (occurring during the last month of pregnancy or within 5 months after delivery)
  * ECG: atrial fibrillation/flutter.
  * Resuscitated sudden death.
  * Early/initial phase of decompensated heart failure.
  * Tamponade complicating pericarditis unless successfully managed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the study's inclusion & exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Value of Heart Rate Lowering Therapy in Acute Myocarditis | baseline
  To study the value of heart rate lowering therapy "pharmacological rest" on the short term in cases of myocarditis without LV dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Hospital, Asyut, Egypt